CLINICAL TRIAL: NCT03155009
Title: An Open-Label, Multicenter, Single-Arm, Phase II Study to Assess the Efficacy and Safety of Alectinib in Patients With ALK-Rearranged Non-Small Cell Lung Cancer After Disease Progression on Prior ALK Inhibitor Therapy
Brief Title: A Study of the Efficacy and Safety of Alectinib in Participants With Anaplastic Lymphoma Kinase (ALK)-Rearranged Non-Small Cell Lung Cancer
Acronym: ATALK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML39349; 2016-003924-22 (EudraCT Number)
Record Dates: First submitted 2017-05-11; First posted 2017-05-16 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — alectinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alectinib (Experimental): 600 mg orally twice daily (BID) for up to 2 years
  Interventions: Drug: Alectinib

INTERVENTIONS:
Drug: Alectinib — 600 mg orally BID with food

SUMMARY:
This study will evaluate the efficacy and safety of alectinib, in selected participants, with anaplastic lymphoma kinase-rearranged (ALK-rearranged) non-small cell lung cancer (NSCLC), after disease progression on prior treatment strategy with crizotinib, as only ALK inhibitor, and eventually chemotherapy treatment(s).

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically or cytologically confirmed locally advanced or metastatic NSCLC (Stage IIIB or IV accordingly to American Joint Committee on Cancer [AJCC] classification)
* Life expectancy of at least 12 weeks, in the opinion of the Investigator
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤ 2
* Having contributive biopsy performed on fresh tissue (FFPE blocks required) taken after progression on previous therapy showing presence of anaplastic lymphoma kinase (ALK) rearrangement, assessed by immunohistochemistry (IHC) and confirmed by fluorescence in situ hybridization (FISH)
* Absence of resistance mechanism to alectinib assessed by the Biomarkers Board
* Disease progression, limited to central nervous system (CNS) without possibility of tissue biopsy
* Non-contributive molecular analyses (not enough tumor cells or deoxyribonucleic acid, [DNA] amount or failure of analyses for technical reasons): inclusion is at investigator discretion (decision made upon Biomarker Board recommendation)
* History of crizotinib exposure
* Washout period: if previous progression on crizotinib: 7 days from last intake of the drug
* If previous progression on chemotherapy: 28 days
* If previous radiation therapy: 15 days
* Participants must have recovered from treatment toxicities to ≤ Grade 1 or to their pretreatment levels (for participants who have developed interstitial lung disease [ILD], they must have fully recovered)
* Recovery from effects of any major surgery, or significant traumatic injury, at least 35 days before the first dose of alectinib
* Adequate hematologic function
* Adequate renal function
* For all females of childbearing potential, a negative pregnancy test must be obtained within three days before starting study drug
* For women who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to remain abstinent or use two adequate methods of contraception, including at least one method with a failure rate of < 1% per year, during the treatment period and for at least 90 days after the last dose of study drug
* For men: agreement to remain abstinent or use a barrier method of contraception (e.g., condom) during the treatment period and for at least 90 days after the last dose of study drug and agreement to refrain from donating sperm during this same period
* Participant has national health insurance coverage

Exclusion Criteria:

* Prior therapy with other ALK inhibitors than crizotinib (including alectinib)
* Participants with symptomatic CNS metastases who are neurologically unstable or require increasing doses of steroids within one week prior to Day 0 to manage CNS symptoms
* Participants with progression limited to CNS and eligible to a focal treatment (surgery or stereotaxic radiotherapy)
* Administration of strong/ potent cytochrome P450 3A (CYP3A) inhibitors or inducers, or agents with potential QT prolonging effects within 14 days prior to first administration of study drug
* Liver disease
* Any clinically significant concomitant disease or condition that could interfere with, or for which the treatment might interfere with, the conduct of the study or the absorption of oral medications or that would, in the opinion of the investigator, pose an unacceptable risk to the participant in this study
* Active or uncontrolled infectious diseases requiring treatment
* History of organ transplant
* Participants with baseline QTc > 470 ms or participants with symptomatic bradycardia
* Pregnant or lactating women
* History of hypersensitivity to any of the additives in the alectinib drug
* Any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol requirements and/or follow-up procedures; those conditions should be discussed with the participant before trial entry
* Serious, uncontrolled infections or current known infection with human immunodeficiency virus (HIV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-09-26 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 2 years
  ORR is defined as the percentage of participants with complete response (CR) or partial response (PR) assessed by the investigator using the Response Evaluation Criteria in Solid Tumors (RECIST), v.1.1. CR is defined as disappearance of all target and non-target lesions and no new lesions, and all pathological lymph nodes must have decreased to <10 mm in short axis. PR is defined as at least a 30% decrease in the sum of diameters of target lesions (taking as reference the baseline sum diameters), no progression in non-target lesions, and no new lesions.

SECONDARY OUTCOMES:
Central Nervous System Objective Response Rate (C-ORR) | Up to 2 years
  C-ORR is defined as the percentage of participants who attain a CR or PR of the baseline CNS metastases based on RECIST v.1.1. CR is defined as disappearance of all target and non-target lesions and no new lesions, and all pathological lymph nodes must have decreased to <10 mm in short axis. PR is defined as at least a 30% decrease in the sum of diameters of target lesions (taking as reference the baseline sum diameters), no progression in non-target lesions, and no new lesions.
Progression-Free Survival (PFS) | Up to 2 years
  PFS is defined as the time between first intake of alectinib and the first occurrence of disease progression, or death from any cause during the study, whichever occurs first. Progressive disease (PD) based on RECIST v.1.1. is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (nadir), including baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time to Progression (TTP) | Up to 2 years
  TTP is defined as the time between first intake of alectinib and the first occurrence of disease progression. PD based on RECIST v.1.1. is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (nadir), including baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Disease Control Rate (DCR) | Up to 2 years
  DCR is defined as the percentage of participants who attain CR, PR, or stable disease (SD) for at least five weeks, based on RECIST v.1.1. CR is defined as disappearance of all target and non-target lesions and no new lesions, and all pathological lymph nodes must have decreased to <10 mm in short axis. PR is defined as at least a 30% decrease in the sum of diameters of target lesions (taking as reference the baseline sum diameters), no progression in non-target lesions, and no new lesions. SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression, taking as reference the smallest sum on study.
Duration of Response (DOR) | Up to 2 years
  DOR is defined as the time from when response (CR or PR), based on RECIST v.1.1, will be first documented to first documented disease progression or death (whichever occurs first). CR is defined as disappearance of all target and non-target lesions and no new lesions, and all pathological lymph nodes must have decreased to <10 mm in short axis. PR is defined as at least a 30% decrease in the sum of diameters of target lesions (taking as reference the baseline sum diameters), no progression in non-target lesions, and no new lesions. PD is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (nadir), including baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Central Nervous System DOR (C-DOR) | Up to 2 years
  C-DOR is defined as the time from the first observation of a CNS response of CR or PR based on RECIST V1.1 until first observation of CNS progression or death from any cause (whichever occurs first). CR is defined as disappearance of all target and non-target lesions and no new lesions, and all pathological lymph nodes must have decreased to <10 mm in short axis. PR is defined as at least a 30% decrease in the sum of diameters of target lesions (taking as reference the baseline sum diameters), no progression in non-target lesions, and no new lesions. PD is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (nadir), including baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Overall Survival (OS) | Up to 2 years
  OS is defined as the percentage of participants alive two years after the start of treatment.
Time to Central Nervous System (CNS) Progression | Up to 2 years
  Time to central nervous system (CNS) progression is defined as the time from first drug intake to first documented occurrence of disease progression in the CNS. PD based on RECIST v.1.1. is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (nadir), including baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Percentage of Participants with Adverse Events (AEs) | Up to 2 years
  An adverse event is considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Preexisting conditions that worsen during the study are reported as adverse events.
Health-Related Quality of Life (QoL), as Assessed by the QLQ-C30 Questionnaire | Up to 2 years
  The QLQ-C30 Questionnaire is used to assess the quality of life of participants with cancer. It includes five functional scales, three symptom scales, a global health status / QoL scale, and six single items. These components range in score from 0 (low response level) to 100 (high response level).
Health-Related QoL, as Assessed by the LC13 Questionnaire | Up to 2 years
  The LC13 Questionnaire includes 13 questions assessing lung cancer-associated symptoms (cough, hemoptysis, dyspnea and site-specific pain), treatment-related side effects (sore mouth, dysphagia, peripheral neuropathy and alopecia), and pain medication. This scale ranges in score from 0 (low response level) to 100 (high response level).
Health-Related QoL, as Assessed by the BN20 Questionnaire | Up to 2 years
  The BN20 Questionnaire includes 20 items assessing future uncertainty, visual disorder, motor dysfunction, communication deficit and other disease symptoms, and treatment toxicities. This scale ranges in score from 0 (low response level) to 100 (high response level).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (16):
- France (16):
  - CHU Angers, Angers
  - Hopital Jean Minjoz; Pneumologie, Besançon
  - Hopital Augustin Morvan; Oncologie Thoracique, Brest
  - Centre Francois Baclesse; Comite 3, Caen
  - Centre Hospitalier Intercommunal; Service de Pneumologie, Créteil
  - Hôpital Nord Michallon; Pneumologie, La Tronche
  - CHRU Lille Service de Pneumologie et Oncologie Thoracique, Lille
  - Hôpital Nord - AP-HM Marseille#, Marseille
  - Hopital Emile Muller;Pneumologie, Mulhouse
  - Institut Curie, Paris
  - Hopital Tenon;Pneumologie, Paris
  - CHU de Bordeaux, Pessac
  - Hopital de Pontchaillou; Service de Pneumologie, Rennes
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen
  - CHU de Toulouse - Hôpital Larrey; Service de pneumologie et oncologie pneumologique, Toulouse
  - Hopital Robert Schuman; Pneumologie, Vantoux